CLINICAL TRIAL: NCT05163938
Title: REThink Chronic-A Mobile Therapeutic Game for the Prevention of Emotional Disorders Among Children Aged 8-16 Years With a Chronic Physical Disease
Brief Title: REThink Chronic-A Mobile Therapeutic Game
Acronym: REThinkChronic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Oana David, Professor, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REThink Chronic
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: REThink Game; Treatment-as-usual
Keywords: chronic physical disease; youth; emotional disorders; therapeutic game; prevention
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: REThink mobile therapeutic game intervention group and Treatment-as-usual group which receives the trial version of the app.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REThink therapeutic game (Experimental): Game based Cognitive-Behavioral Therapy: REThink therapeutic game is an online therapeutic game developed by David and collaborators (2018).
  The seven levels of the game were developed based on the REBT model and each level trains an ability:
  Level 1: identify the emotional reactions, and differentiating between basic emotions, complex emotions, and functional and dysfunctional emotions; Level 2: identify cognitive processes.
  Level 3: identify the relation between cognitive processes, emotions, and behavioral reactions; Level 4: change irrational cognitions into rational cognitions; Level 5: build problem-solving skills; Level 6: build relaxation skills; Level 7: consolidate of the previous skills and building happiness skills. A new level will be unlocked once every three days. In order for a level to be unlocked, the previous one must have been completed.
  Duration of the intervention: 21 days (a total of seven levels unlocked every three days)
  Interventions: Device: REThink Therapeutic Game
- Treatment as usual (Active Comparator): In the treatment as usual group the child/adolescent benefits from a free trial version of the REThink game which means a shorter version of each level of the game.
  Interventions: Device: Treatment as Usual

INTERVENTIONS:
Device: REThink Therapeutic Game — Game based Cognitive-Behavioral Therapy: REThink therapeutic game is an online therapeutic game developed by David and collaborators (2018).
  The seven levels of the game were developed based on the REBT model and each level trains an ability:
  Level 1: identify the emotional reactions, and differentiating between basic emotions, complex emotions, and functional and dysfunctional emotions; Level 2: identify cognitive processes.
  Level 3: identify the relation between cognitive processes, emotions, and behavioral reactions; Level 4: change irrational cognitions into rational cognitions; Level 5: build problem-solving skills; Level 6: build relaxation skills; Level 7: consolidate of the previous skills and building happiness skills. A new level will be unlocked once every three days. In order for a level to be unlocked, the previous one must have been completed.
  Duration of the intervention: 21 days (a total of seven levels unlocked every three days)
  Arms: REThink therapeutic game
Device: Treatment as Usual — Treatment As Usual: In the treatment as usual group the child/adolescent benefits from a free trial version of the REThink game which means a shorter version of each level of the game.
  Arms: Treatment as usual

SUMMARY:
The general objective of the study is to test the efficacy of an online therapeutic game (REThink Game) for the prevention of emotional disorders in children and adolescents aged between 8-16 years with a chronic physical disease.

DETAILED DESCRIPTION:
The objective of the study is to test an online therapeutic game which, being an evidence-based prevention tool for children and adolescents, might contribute to preventing emotional disorders in children and adolescents aged between 8-16 years old diagnosed with a chronic physical disease. REThink is a scientifically validated therapeutic game for children and adolescents to improve their emotional skills. The enrollment will take place both online and in pediatric medical institutions. The research study will include one parent of the eligible child/adolescent. The children and adolescents will be randomized into two equal groups: the intervention group which benefits of the entire REThink game and the treatment-as-usual group which benefits of a free trial version of the app. Three assessments will be performed to evaluate the variables of interest: before intervention (baseline), after intervention (post-intervention), and a follow-up six months after the post-intervention assessment was performed.

ELIGIBILITY:
Inclusion Criteria:

* are aged 8 to 16 years old
* are diagnosed with a chronic physical disease
* have consent from the parent or legal tutor to participate in the study
* are fluent in Romanian
* have access to a mobile phone, tablet or laptop

Exclusion Criteria:

* have intellectual disabilities or physical limitations which make it impossible for the them to play the game
* have traumatic brain injuries
* have a diagnosed mental disorder
* demised during the study period

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Children's emotional symptoms | 7 months
  The Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997; Goodman et al.,1998)
Children's negative and positive affect | 7 months
  The Positive and Negative Affect Schedule (PANAS-C; Laurent et al, 1999)

SECONDARY OUTCOMES:
Child emotion regulation | 7 months
  The Cognitive Emotion Regulation Scale (CERQ-K; Orgilés, 2017) aims to identify the emotional cognitive regulation strategies that a child uses after going through negative or stressful events.
Children's irrational beliefs | 7 months
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/ rational beliefs as a mechanism of change.
Children's quality of life | 7 months
  Youth Quality of Life Instrument - Short Form (YQOL-SF- Edwards, Huebner, Connell & Patrick, 2002; Patrick, Edwards & Topolski, 2002) is a questionnaire which assesses the general quality of life in children and adolescents aged 11 to 18 years old with and without chronic diseases and disabilities. The short form consists of 15 items which evaluate the domains of sense of self, social relationships, environment, and general quality of life.
Emotional state | 7 months
  MoodWheel (MoodWheel; David, 2016) is a web and mobile application that includes procedures for sampling experience in order to assess present/past emotional difficulties, as well as positive emotions. The purpose of the mobile app is to examine the validity, control and functionality of the emotion felt by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Oana David, PhD, Study Director — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No